CLINICAL TRIAL: NCT02286336
Title: The Minimum Effective Concentration of Ropivacaine in Ultrasound-guided Supraclavicular Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Fang Gang, Dr., Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-64
Record Dates: First submitted 2014-11-02; First posted 2014-11-07 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Minimum Effective Concentration of Local Anesthetic
Keywords: minimum effective concentration; ropivacaine; ultrasound-guided supraclavicular block
MeSH Terms: interventions — Brachial Plexus Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- middle aged group (Experimental): brachial plexus block with ropivacaine 40ml, MEC90 for USG-SCB
  Interventions: Other: brachial plexus block
- young group (Active Comparator): brachial plexus block with ropivacaine 40ml, MEC90 for USG-SCB
  Interventions: Other: brachial plexus block

INTERVENTIONS:
Other: brachial plexus block — brachial plexus block with ropivacaine 40ml
  Other Names: ultrasound guided supraclavicular block

SUMMARY:
The aim of this study is to determine the minimum effective concentration of local anesthetic (ropivacaine 40mL) required to produce an effective double-injection USG-SCB for surgical anesthesia in 90% of patients (MEC90) in young group (18-40 years) and in middle aged group (40-65 years) of patients scheduled for elective surgery of one upper limb distal to the shoulder.

DETAILED DESCRIPTION:
The study is based on biased coin design, and the concentration of LA for the next patient is determined by the result of the last one. In the case of block failure, the concentration will be increased by 0.025%. Conversely, block success will result in either a reduction in concentration by 0.025% (probability 11%) or no change in concentration (probability 89%). A blinded assistant will assess sensory and motor blockade in each nerve territory ( the median, radial, ulnar and musculocutaneous nerves) at 10-min intervals up to 30 min after completion of the block. Finally, MEC90 is calculated by isotonic regression.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years
2. ASA 1-3
3. body mass index between 18 and 35kg/m2

Exclusion Criteria:

1. inability to consent to the study
2. pregnancy
3. allergy to local anesthetics
4. preexisting neuropathy or coagulopathy
5. prior surgery in the supraclavicular region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The Minimum Effective Concentration of Ropivacaine in Ultrasound-guided Supraclavicular Block | up to 6 months
  The Minimum Effective Concentration (MEC) of Ropivacaine in Ultrasound-guided Supraclavicular Block is based on 60 measurements in 60 patients (secondary outcome measure: block success). MEC is determined by biased coin design method when all patients have been tested in the study.

SECONDARY OUTCOMES:
Block success | up to 30 minutes after nerve block is performed
  A blinded Assistant assess the sensory and motor block onset time for each nerve (median, radial, ulnar and musculocutaneous) at 10-min intervals up to 30 min after completion of the block.

CONTACTS AND LOCATIONS:
Overall Officials: Ailin Luo, MD.,PhD, Study Chair — Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China